CLINICAL TRIAL: NCT00195988
Title: Comparison Of Efficacy Of Two Immunosuppressive Protocols Including Tacrolimus With Or Without Mycophenolate Mofetil In Pediatric Liver Transplantation Aimed In Early Termination Of Steroid Therapy
Brief Title: Comparison of Immunosuppression Protocols After LTx in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Memorial Health Institute, Poland (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDS-CZD-piokal
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-11-17 (Estimated); Status verified 2005-06

CONDITIONS: Liver Transplantation
Keywords: immunosuppression,; steroid avoidance,; liver transplantation,; children
MeSH Terms: interventions — Tacrolimus; Steroids; Mycophenolic Acid

INTERVENTIONS:
Drug: tacrolimus, steroids, mycophenolate mofetil

SUMMARY:
Open label, randomised, prospective, onecentre Investigator Driven Study:

Comparison of two protocols of immunosuppression after liver Tx in children:

A: Study group - FK506-MMF. Immunosupression protocol: Methylprednisolone 10 mg/kg intraoperatively i.v. FK506 Day 0 or 1 orally (0,15 mg/kg/D in two doses).MMF max. dosage 30 mg/kg/D p.o. day 0 through day 90.

B. Control group - Tacrolimus, steroids. Immunosupression protocol: Methylprednisolone 10 mg/kg bm intraoperatively Children < 25kg bm: Methylprednisolone taper from 100 mg/D on day 0 to MP 10 mg on day 7 Children > 25kg bm: Methylprednisolone taper from 200 mg/D on day 0 to MP 20 mg on day 7 Week 2-4 Prednisone - 0,5-0,3 mg/kg/D; Week 4-12 Prednisone -0,3-0,2 mg/kg/D; Month 4-6 Prednisone 0,2 - 0,1 mg/kg/D Month 7 - Steroid withdrawal FK506 Day 0 or 1 orally (0,15 mg/kg/D in two doses).

Primary end points:

Number of rejections, number of steroid-resistant rejections.

Secondary end points:

Patients and graft survival Dyslipidemia one year after transplantation Hypertension one year after transplantation Hyperglycemia/Diabetes de novo one year after transplantation Renal function before Tx and 1 year after Tx

DETAILED DESCRIPTION:
A: Study group

FK506-MMF.

Immunosupression protocol:

Metylprednisolon 10 mg/kg intraoperatively i.v.

FK506 Day 0 or 1 oraly (0,15 mg/kg/D in two doses).

MMF max. dosage 30 mg/kg/D p.o. day 0 through day 90 according to patient condition and therapeutic MMF blood concentration

Tailoring:

Immunosupression protocol will be tailored according to the cause of liver failure: patients with autoimmune liver disease (autoimmune hepatitis, PBC, PSC, overlap syndrome etc) would be maintained on MMF. All other recipients including cryptogenic liver cirrhosis will be gradually (over 1 month) withdrawn from MMF administration 90 days after transplantation if there is:

1. good kidney function (S-creatinin < 150 umol/l) enabling to achieve and maintain Tacrolimus trough levels above 6 ng/ml and
2. if there was no more than one episode of acute rejection of the graft which resolved completely.

Targeted Tacrolimus trough levels:

Month 1 - 3 through levels 10-15 ng/ml Month 4-6 10-12 ng/ml Month 7-12 10 - 6 ng/ml

Rejection treatment:

1. Tacrolimus dose adjustment to upper limit of target level if last Tacrolimus trough level is below the intended limit.
2. Steroid boluses would be administered Metylprednisolon 10 mg/kg daily 3 consecutive days. No steroid taper. Control biopsy after normalisation of LFTs.
3. After two attacks of acute rejection before MMF disontinuation Prednison dose would be introduced on at least 0,3 mg/D for 3 months.
4. After second attack of AR after MMF discontinuation Prednison dose would be introduced on at least 0,3 mg/D for 6 months.
5. Steroid resistant rejection: biopsy proven rejection persisting after three courses of steroid pulses. Steroid resistant rejection would be treated according to local praxis.

Concomitant drugs:

Antiviral and antibacterial prophylaxis according to current centre praxis. Prophylaxis of cholestasis and prophylaxis/treatment of the bone disease where applicable.

B. Control group

Tacrolimus, steroids.

Immunosupression protocol:

Metylprednisolon 10 mg/kg bm intraoperatively Children < 25kg bm: Metylprednisolon taper from 100 mg/D on day 0 to MP 10 mg on day 7 Children > 25kg bm: Metylprednisolon taper from 200 mg/D on day 0 to MP 20 mg on day 7 Week 2-4 Prednison - 0,5-0,3 mg/kg/D Week 4-12 Prednison -0,3-0,2 mg/kg/D Month 4-6 Prednison 0,2 - 0,1 mg/kg/D Month 7 - Steroid withdrawal

FK506 Day 0 or 1 orally (0,15 mg/kg/D in two doses).

Intended Tacrolimus trough levels:

Month 1 -3 through levels 10-15 ng/ml Month 4-6 10-12 ng/ml Month 7-12 6-10 ng/ml

Rejection treatment:

1. Tacrolimus dose adjustment to upper limit of target level if last Tacrolimus trough level is below the intended limit.
2. Steroid boluses would be administered Metylprednisolon 10 mg/kg bm daily 3 consecutive days. No steroid taper, return to previous steroid dose. Control biopsy after normalisation of LFTs.
3. After two attacks of acute rejection Prednison dose would be maintained on at least 0,3 mg/D for 3 months.
4. Steroid resistant rejection: biopsy proven rejection persisting after three courses of steroid pulses. Steroid resistant rejection would be treated according to local praxis.

Biopsy: Liver biopsy should be taken in any suspicion of graft rejection or disease recurrence. Protocol biopsy would be taken according to local practice, liver biopsy in one-year after transplantation is mandatory.

Primary end points:

Number of rejections, number of steroid-resistant rejections.

Secondary end points:

Patients and graft survival Dyslipidemia one year after transplantation Hypertension one year after transplantation Hyperglycemia/Diabetes de novo one year after transplantation Renal function before Tx and 1 year after Tx

Inclusion criteria:

Subjects who meet all of the following criteria are eligible for this study:

1. Male or female patients, not older than 18 years old.
2. Primary liver transplantation
3. Patient is capable of understanding the purpose and risks of the study and has been informed both orally and in writing and has given informed consent

Exclusion criteria:

Subjects who meet one or more of the following criteria are not eligible for this study:

1. Female patients who are pregnant or are breast feeding
2. Patients > 18 years old
3. Combined liver-kidney transplantation
4. Recipient of second liver graft
5. Patients are allergic, hyper-sensitive or intolerant to HCO-60 or structurally related compounds, macrolide antibiotics or tacrolimus.
6. Patients with known HIV-anamnesis
7. Patient requires ongoing dosing with a systemic immunosuppressive drug at study entry for another indication than the prophylaxis of liver graft rejection
8. Patient has significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, or active peptic ulcer.
9. Patient is participating or has participated in another clinical study and/or is taking or has been taking an investigational drug in the past 28 days.
10. Other reasons which depend on the assessment of the physician (no MMF will be given to patients with severe persistent hypersplenism (WBC < 3.500/ml, platelets < 50.000/ml)

Informed Consent:

Patient, who will give written consent for participation in the study and will fulfil all the inclusion and exclusion criteria, will be included in the study. After inclusion into the study, the patient may withdraw at any time for any reason.

Follow-up: (time of one patient observation ) -12 months

Number of centers: 1 Number of patients: 40 Indication: - Primary Liver transplantation Duration of study: 36 months Enrollment period: 18 months

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria are eligible for this study:

  1. Male or female patients, not older than 18 years old.
  2. Primary liver transplantation
  3. Patient is capable of understanding the purpose and risks of the study and has been informed both orally and in writing and has given informed consent

Exclusion Criteria:

* Subjects who meet one or more of the following criteria are not eligible for this study:

  1. Female patients who are pregnant or are breast feeding
  2. Patients > 18 years old
  3. Combined liver-kidney transplantation
  4. Recipient of second liver graft
  5. Patients are allergic, hyper-sensitive or intolerant to HCO-60 or structurally related compounds, macrolide antibiotics or tacrolimus.
  6. Patients with known HIV-anamnesis
  7. Patient requires ongoing dosing with a systemic immunosuppressive drug at study entry for another indication than the prophylaxis of liver graft rejection
  8. Patient has significant, uncontrolled concomitant infections and/or severe diarrhoea, vomiting, or active peptic ulcer.
  9. Patient is participating or has participated in another clinical study and/or is taking or has been taking an investigational drug in the past 28 days.
  10. Other reasons which depend on the assessment of the physician (no MMF will be given to patients with severe persistent hypersplenism (WBC < 3.500/ml, platelets < 50.000/ml)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2002-09; Study Completion 2006-07

PRIMARY OUTCOMES:
Number of rejections, number of steroid-resistant rejections.

SECONDARY OUTCOMES:
Patients and graft survival
Dyslipidemia one year after transplantation
Hypertension one year after transplantation
Hyperglycemia/Diabetes de novo one year after transplantation
Renal function before Tx and 1 year after Tx

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kalicinski, Prof., MD, PhD, Principal Investigator — Children's Memorial Health Institute
Locations (1):
- Department of Pediatric Surgery and Organ Transplantation, CMHI, Warsaw, Poland